CLINICAL TRIAL: NCT03240445
Title: A Part-randomised, Single Centre, Single Dose, Crossover,Phase I Study to Investigate the Impact of Changes to the Dosing Regimen on the Pharmacokinetic Profile of ODM-203 in Healthy Male Volunteers
Brief Title: Impact of Changing the Dosing Regimen on the PK Profile of ODM-203
Acronym: KIPEV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Collaborators: Quotient Clinical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 3113004
Record Dates: First submitted 2017-07-26; First posted 2017-08-07 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Period 1 (Experimental): ODM-203 dosed after food
  Interventions: Drug: ODM-203 (Period 1)
- Period 2 (Experimental): ODM-203 dosed before food
  Interventions: Drug: ODM-203 (Period 2)
- Periods 3-6 (Experimental): ODM-203 dosed as a tablet or dispersion
  Interventions: Drug: ODM-203 (Periods 3-6)

INTERVENTIONS:
Drug: ODM-203 (Period 1) — ODM-203 400mg as tablets taken 30 minutes after food
  Arms: Period 1
Drug: ODM-203 (Period 2) — ODM-203 400mg as tablets taken 1 hour before a light breakfast
  Arms: Period 2
Drug: ODM-203 (Periods 3-6) — ODM- 203 400mg as tablets for oral administration or 400mg as oral dispersion either before/after food
  Arms: Periods 3-6

SUMMARY:
This Phase I study in healthy male volunteers will evaluate the impact of the effect of food on the pharmacokinetic profile of ODM-203.

DETAILED DESCRIPTION:
This study will be a single dose part randomised cross over study with up to 6 study periods. ODM-203 may be dosed using a variety of different conditions with respect to food depending on emerging data. The impact of changing the presentation of ODM-203 may also be assessed to determine the PK of alternative formulations and identify appropriate drug formulations for further development.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Able to speak, write and understand English
* Body mass index of 18.0-32.0
* Weight 55-95 kg
* Adequate method of contraception
* Good state of health

Exclusion Criteria:

* Receipt of IMP in a clinical research study or donation/loss of >400ml blood within previous 3 months or previously enrolled in this study
* History of drug or alcohol abuse or positive drugs of abuse test or regular alcohol consumption or current smoker/user of nicotine replacement products
* Positive drugs of abuse test
* Positive hepatitis B, hepatitis C or HIV results
* Donation/loss of >400ml blood within previous 3 months
* Poor compliance or inability to follow protocol requirements/instructions/restrictions.
* Vulnerable subjects
* Evidence of clinically relevant disease of any body system including relevant psychiatric disorders or conditions requiring regular concomitant medication
* History of significant hypersensitivity, anaphylaxis, intolerance to drugs/food
* Propensity to get headaches when refraining from caffeine containing beverages
* Any abnormal laboratory value, vital signs, ECG parameter or physical examination interfering with the test results or causing a health risk for the subject or failure to satisfy the investigator of fitness to participate for any other reason.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy male
Enrollment: 16 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2017-10-23 (Actual); Study Completion 2017-10-23 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration curve(AUC) ODM-203 in the presence and absence of food | 0 to 72 hours
  Area under the plasma concentration curve (AUC) will be measured to investigate the pharmacokinetic profile of ODM-203 in the presence and absence of food

SECONDARY OUTCOMES:
Number of adverse events | From the date of informed consent to the date of the end of study estimated to be up to 17 weeks
  Number of adverse events counts
Area under the plasma concentration curve(AUC) ORM-21444 in the presence and absence of food | 0 to 72 hours
  Area under the plasma concentration curve (AUC) will be measured to investigate the pharmacokinetic profile of ORM-21444 in the presence and absence of food

CONTACTS AND LOCATIONS:
Overall Officials: Clare Preskey, BSc, Study Director — Quotient Clinical
Locations (1):
- Quotient Clinical Ltd, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided